CLINICAL TRIAL: NCT04048382
Title: Developing a Patient Navigation Intervention for PrEP Continuum of Care Among Young Latino MSM (PrEParate)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Blashill, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-2017-0187; 1R34MH114699-01 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: HIV/AIDS
Keywords: HIV Seroprevalence; Pre-Exposure Prophylaxis; Patient Navigation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation (PN) (Experimental): This intervention consists of standardized health educational materials and manualized sessions that can be implemented based on a participant's stage in the PrEP continuum. The intervention will utilize bilingual peer lay navigators and also consist of barrier reduction strategies to assist individuals with implementing HIV prevention, including the use of PrEP.
  Interventions: Behavioral: Patient Navigation
- Usual Care (UC) (Other): Participants in this condition will receive the CDC's 2-page PrEP Information Sheet in the participant's preferred language (either English or Spanish).
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Patient Navigation — Spanish-English bilingual peer lay navigators hired by Family Health Centers of San Diego will provide the PN intervention during the study, trained using manuals developed in formative research and via the Patient Navigation Research Program training approach. Services will generally focus on: 1) overcoming community, health system, interpersonal, and individual barriers to accessing PrEP-related healthcare; 2) increasing each patient's knowledge, attitudes, and self-efficacy for initiating and adhering to PrEP; 3) improving communication between the patient and healthcare team through appointment scheduling and reminders; and 4) sexual risk reduction counseling.
  Arms: Patient Navigation (PN)
Other: Usual Care — The booklet given is a 2-page booklet including the following information: 1) overview of PrEP; 2) eligibility for PrEP; 3) efficacy of PrEP; 4) safety of PrEP; and 5) obtaining, initiating, and adhering to PrEP. Participants will also be provided with both verbal and written information regarding available sexual health and HIV prevention services, including PrEP, at Family Health Centers of San Diego (FHCSD). Comprehensive HIV-prevention healthcare, including PrEP, is available to study participants at FHCSD at no or minimal cost. If a UC participant is diagnosed with a sexually transmitted infection, including HIV, treatment and follow-up will be coordinated by FHCSD staff as per usual care procedures.
  Arms: Usual Care (UC)

SUMMARY:
This study aims to help young Latino gay and bisexual men access sexual health information, including PrEP. Participants will be randomly assigned to either the patient navigation or the usual care condition and followed for 6 months. The study will recruit self-identified Latino men between the ages of 18 and 29 who also identify as gay, bisexual, and/or have sex with other men, and report CDC defined HIV risk behaviors.

DETAILED DESCRIPTION:
Reducing the number of new human immunodeficiency virus (HIV) infections is one of the goals of the National HIV/AIDS Strategy and an objective of Healthy People 2020. Men who have sex with men (MSM) are the most at risk group for contracting HIV in the U.S., comprising 67% of the total new HIV diagnoses in 2014. The HIV epidemic impacts some groups of MSM disproportionately, with Latino MSM comprising 25.1% of new HIV infections among MSM between the ages of 13 and 29 years. Moreover, between 2010 and 2014, incidence of HIV increased 13% among Latino MSM, while all other racial/ethnic MSM groups showed stable or decreasing trends, underscoring the vulnerability of HIV infection among Latino MSM.

Pre-exposure prophylaxis (PrEP), a medication taken daily to reduce risk of becoming infected with HIV, was approved by the Food and Drug Administration (FDA) in 2012, and has demonstrated strong efficacy. When taken consistently, PrEP has been shown to reduce new incidence of HIV by 92%. Despite the promise of PrEP to transform HIV prevention, there remain significant barriers to PrEP use among those who would benefit the most, including low awareness, knowledge, medical mistrust, perceived high costs, lack of access, language barriers, low health literacy, and stigma. In a recent study conducted among 600 MSM between the ages of 18 and 29 years in Southern California, Latino MSM reported the lowest levels of use at 6.6%, compared to 9.8% and 13.9% for Black and White participants, respectively. Although Latino MSM reported the lowest use of PrEP, they also reported the greatest willingness to use PrEP compared to White and Black MSM. This discrepancy in willingness versus actual PrEP use among Latino MSM emphasizes the need to intervene to address barriers among this population.

There are a number of different steps that individuals must take to initiate, regularly adhere to, and persist in taking PrEP, with each step in this cascade associated with its own unique barriers. One approach that has been used to address multiple barriers to adhering to recommended health care is patient navigation (PN). PN has been successfully utilized to facilitate access to healthcare among other Latino populations and peer PN may be an ideal intervention to aid in PrEP uptake among Latino MSM by assisting individuals in overcoming barriers to obtaining and using PrEP. To our knowledge, no known PN programs for PrEP have been developed or pilot tested specifically for Latino MSM.

The proposed study will engage young Latino MSM, a population at substantial risk for HIV infection, to pilot-test a peer PN intervention designed to improve engagement and retention in PrEP care. The peer PN intervention will be pilot-tested by comparing it to receipt of usual medical care (UC) plus written information. Individuals randomized to PN will receive the services of a peer patient navigator who will collaborate with the patient, his partner(s), health care professionals, and support service professionals to improve awareness of PrEP, facilitate engagement and retention in PrEP care, and provide strategies for adherence to PrEP. PN will be compared to UC at a 3 and 6-month follow-ups to evaluate the acceptability and feasibility of the PN intervention, and the preliminary impact of the PN intervention on engagement in PrEP-related care and PrEP adherence. In response to RFA-MH-17-361 "Improving the HIV PrEP Cascade-R34," the investigators propose:

To conduct a pilot randomized controlled trial of the patient navigation intervention by comparing it to usual care to assess feasibility, acceptability, and preliminary impact. The investigators plan to randomize 60 young Latino MSM participants to either the PN or UC condition and follow participants for 6 months. It is expected that the pilot test will provide information about the feasibility and acceptability of the intervention and study methods, in preparation for a future full-scale efficacy trial. In addition, the pilot test will evaluate its preliminary impact on 7 PrEP cascade-related outcomes (i.e., scheduled and attended PrEP consultation; PrEP prescription received; PrEP prescription filled; PrEP initiated; self-reported PrEP adherence; and PrEP follow-up medical appointment attended).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 29 years
2. Identifies as male
3. Identifies as gay/bisexual or reports having sex with men in past 12 months
4. Identifies as Latino/Hispanic
5. Self-reports being HIV-uninfected
6. Resides in San Diego County, California
7. Speaks English or Spanish
8. Willing and able to provide informed consent
9. Willing to receive PrEP-related health care at FHCSD
10. Reports at least one HIV risk factor as informed by CDC guidelines

10a. MSM are at elevated risk for HIV (as per CDC) if they report one of the following:

* an HIV-infected sexual partner
* diagnosis of a bacterial STI within the past 12 months
* engaging in condomless anal sex with a non-monogamous partner in the past 12 months
* engaging in commercial sex work in the past 12 months
* injection of illicit drugs and sharing of injection equipment in the past 12 months
* engaging in drug treatment for injection drug use in the past 12 months.

Exclusion criteria:

1. HIV-infected

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity. The relevant eligibility question is, "Do you identify as male?"
Enrollment: 57 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Blashill, PhD, Principal Investigator — San Diego State University; Kristen Wells, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith DK, Van Handel M, Wolitski RJ, Stryker JE, Hall HI, Prejean J, Koenig LJ, Valleroy LA. Vital Signs: Estimated Percentages and Numbers of Adults with Indications for Preexposure Prophylaxis to Prevent HIV Acquisition--United States, 2015. MMWR Morb Mortal Wkly Rep. 2015 Nov 27;64(46):1291-5. doi: 10.15585/mmwr.mm6446a4. PMID 26606148
- [Background] Anderson PL, Glidden DV, Liu A, Buchbinder S, Lama JR, Guanira JV, McMahan V, Bushman LR, Casapia M, Montoya-Herrera O, Veloso VG, Mayer KH, Chariyalertsak S, Schechter M, Bekker LG, Kallas EG, Grant RM; iPrEx Study Team. Emtricitabine-tenofovir concentrations and pre-exposure prophylaxis efficacy in men who have sex with men. Sci Transl Med. 2012 Sep 12;4(151):151ra125. doi: 10.1126/scitranslmed.3004006. PMID 22972843
- [Background] Calhoun EA, Whitley EM, Esparza A, Ness E, Greene A, Garcia R, Valverde PA. A national patient navigator training program. Health Promot Pract. 2010 Mar;11(2):205-15. doi: 10.1177/1524839908323521. Epub 2008 Dec 30. PMID 19116415
- [Background] Jean-Pierre P, Fiscella K, Winters PC, Post D, Wells KJ, McKoy JM, Battaglia T, Simon MA, Kilbourn K; Patient Navigation Research Program Group. Psychometric development and reliability analysis of a patient satisfaction with interpersonal relationship with navigator measure: a multi-site patient navigation research program study. Psychooncology. 2012 Sep;21(9):986-92. doi: 10.1002/pon.2002. Epub 2011 Jun 17. PMID 21681995
- [Background] Katz ML, Young GS, Reiter PL, Battaglia TA, Wells KJ, Sanders M, Simon M, Dudley DJ, Patierno SR, Paskett ED. Barriers reported among patients with breast and cervical abnormalities in the patient navigation research program: impact on timely care. Womens Health Issues. 2014 Jan-Feb;24(1):e155-62. doi: 10.1016/j.whi.2013.10.010. PMID 24439942
- [Background] Centers for Disease Control and Prevention. Diagnoses of HIV infection in the United States and dependent areas, 2014. HIV Surveillance Report. 2015;26:1-123.
- [Background] Pulsipher CA MJ, Plant A, Curtis P, Holloway IW, Leibowitz AA. Addressing PrEP Dispartities Among Young Gay and Bisexual Men in California. California HIV/AIDS Research Program, 2016 September. Report No.
- [Background] Golub SA, Gamarel KE, Rendina HJ, Surace A, Lelutiu-Weinberger CL. From efficacy to effectiveness: facilitators and barriers to PrEP acceptability and motivations for adherence among MSM and transgender women in New York City. AIDS Patient Care STDS. 2013 Apr;27(4):248-54. doi: 10.1089/apc.2012.0419. PMID 23565928
- [Background] Bauermeister JA, Meanley S, Pingel E, Soler JH, Harper GW. PrEP awareness and perceived barriers among single young men who have sex with men. Curr HIV Res. 2013 Oct;11(7):520-7. doi: 10.2174/1570162x12666140129100411. PMID 24476355
- [Background] Ayala G, Makofane K, Santos GM, Beck J, Do TD, Hebert P, Wilson PA, Pyun T, Arreola S. Access to Basic HIV-Related Services and PrEP Acceptability among Men Who Have sex with Men Worldwide: Barriers, Facilitators, and Implications for Combination Prevention. J Sex Transm Dis. 2013;2013:953123. doi: 10.1155/2013/953123. Epub 2013 Jul 8. PMID 26316968
- [Background] Lui A, Colfax G, Cohen S, Bacon O, Kolber M, Amico K, et al., editors. The spectrum of engagement in HIV prevention: Proposal for a PrEP cascade. 7th International conference on HIV treatment and prevention adherence; 2012; Miami Beach, Florida.
- [Background] Braschi CD, Sly JR, Singh S, Villagra C, Jandorf L. Increasing colonoscopy screening for Latino Americans through a patient navigation model: a randomized clinical trial. J Immigr Minor Health. 2014 Oct;16(5):934-40. doi: 10.1007/s10903-013-9848-y. PMID 23736964
- [Background] Enard KR, Nevarez L, Hernandez M, Hovick SR, Moguel MR, Hajek RA, Blinka CE, Jones LA, Torres-Vigil I. Patient navigation to increase colorectal cancer screening among Latino Medicare enrollees: a randomized controlled trial. Cancer Causes Control. 2015 Sep;26(9):1351-9. doi: 10.1007/s10552-015-0620-6. Epub 2015 Jun 25. PMID 26109462
- [Background] Wilson FA, Villarreal R, Stimpson JP, Pagan JA. Cost-effectiveness analysis of a colonoscopy screening navigator program designed for Hispanic men. J Cancer Educ. 2015 Jun;30(2):260-7. doi: 10.1007/s13187-014-0718-7. PMID 25168070
- [Background] Medsharing I. Randomizer for Clinical Trial. Fontenay Sous Bois, France: Medsharing, Inc.; 2016.
- [Background] Bartholomew LK, Parcel GS, Kok G, Gottlieb NH, Fernandez ME. Planning health promotion programs: An intervention mapping approach. Third ed. San Francisco, California: Jossey-Bass; 2011
- [Background] Attkisson CC, Greenfield TK. The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In: Maruish ME, editor. The use of psychological testing for treatment planning and outcomes assessment. 3. 3rd ed. Mahwah, New Jersey: Lawrence Erlbaum Associates; 2004
- [Background] McKenna SP, Doward LC. The translation and cultural adaptation of patient-reported outcome measures. Value Health. 2005 Mar-Apr;8(2):89-91. doi: 10.1111/j.1524-4733.2005.08203.x. No abstract available. PMID 15804316
- [Background] Swaine-Verdier A, Doward LC, Hagell P, Thorsen H, McKenna SP. Adapting quality of life instruments. Value Health. 2004 Sep-Oct;7 Suppl 1:S27-30. doi: 10.1111/j.1524-4733.2004.7s107.x. PMID 15367241
- [Background] Epstein J, Santo RM, Guillemin F. A review of guidelines for cross-cultural adaptation of questionnaires could not bring out a consensus. J Clin Epidemiol. 2015 Apr;68(4):435-41. doi: 10.1016/j.jclinepi.2014.11.021. Epub 2014 Dec 17. PMID 25698408
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Knodel J. The design and analysis of focus group studies: A practical approach. Successful focus groups: Advancing the state of the art. 1. London: Sage Publications; 1993. p. 35-50.
- [Background] Inc. SI. SAS software version 9.4. Cary, NC: SAS Institute; 2013.
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Derived] Blashill AJ, Gordon JR, Rojas SA, Ramers CB, Lin CD, Carrizosa CM, Nogg KA, Lamb KM, Lucido NC, Jones IJ, Rivera D, Cobian Aguilar RA, Brady JP, Fuentes M, Wells KJ. Pilot randomised controlled trial of a patient navigation intervention to enhance engagement in the PrEP continuum among young Latino MSM: a protocol paper. BMJ Open. 2021 May 26;11(5):e040955. doi: 10.1136/bmjopen-2020-040955. PMID 34039570
- See also: Family Health Centers of San Diego. LGBT services 2015 [cited 2019 February 22]. — http://www.fhcsd.org/lgbt-services
- See also: United States Census Bureau. QuickFacts: San Diego County, California; California 2019 [April 13, 2019]. — http://www.census.gov/quickfacts/fact/table/sandiegocountycalifornia,ca/PST045218
- See also: Newport F, Gates G. San Francisco Metro Area Ranks Highest in LGBT Percentage 2015 [cited 2016 June 1]. — http://www.gallup.com/poll/182051/san-francisco-metro-area-ranks-highest-lgbt-percentage.aspx
- See also: US Public Health Service. Preexposure Prophylaxis for the Prevention of HIV infection in the United States-2014 Clinical Practice Guideline 2014 [cited 2017 January 5]. — http://www.cdc.gov/hiv
- See also: Family Health Centers of San Diego. Welcome to gay men's health service 2015 [February 11, 2019]. — http://gaymenshealth.org

RESULTS

PARTICIPANT FLOW:
Period: 3-Month Follow Up
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Started | 28 | 29
Completed | 26 | 28
Not Completed | 2 | 1
Not completed — Enrolled but did not complete survey | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: 6-Month Follow up
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Started | 28 | 28
Completed | 26 | 28
Not Completed | 2 | 0
Not completed — Enrolled but did not complete survey | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Navigation (PN) | Usual Care (UC) | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.07 (2.45) | 25.59 (3.01) | 25.33 (2.73)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Categorical data was collected on sex/gender.
  Participants
    Male | 24 | 27 | 51
    Non-binary | 3 | 2 | 5
    Transgender | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 29 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 28 | 29 | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants That Scheduled an Appointment for PrEP Consultation.
Description: Participants will be asked if they have scheduled an appointment for PrEP consultation on a follow up questionnaire. It will be confirmed by reviewing their medical records.
Time Frame: 3 months
Population: Number of participants analyzed= 53 due to missing data. This question was displayed contingent on answering "Yes" to "Before this study, had you ever heard of PrEP?"
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Number analyzed (Participants) | 26 | 27
Participants | 10 | 11
Statistical Analysis 1: Comparison: Patient Navigation (PN) vs Usual Care (UC); Test type: Superiority; p = .88, Regression, Logistic; Odds Ratio (OR) = 1.1

2. Primary Outcome: Percent of Participants That Attended an Appointment for PrEP Consultation.
Description: Participants will be asked if they have attended an appointment for PrEP consultation on a follow up questionnaire. It will be confirmed by reviewing their medical records.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Number analyzed (Participants) | 26 | 27
Participants | 10 | 11
Statistical Analysis 1: Comparison: Patient Navigation (PN) vs Usual Care (UC); Test type: Superiority; p = .49, Regression, Logistic; Odds Ratio (OR) = 1.7

3. Primary Outcome: Percent of Participants That Received a PrEP Prescription.
Description: Participants will be asked if they have received a PrEP prescription on a follow up questionnaire. It will be confirmed by reviewing their medical records.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Number analyzed (Participants) | 26 | 27
Participants | 12 | 12
Statistical Analysis 1: Comparison: Patient Navigation (PN) vs Usual Care (UC); Test type: Superiority; p = .91, Regression, Logistic; Odds Ratio (OR) = 1.1

4. Primary Outcome: Percent of Participants That Filled Their PrEP Prescription.
Description: Participants will be asked if they have filled their PrEP prescription on a follow up questionnaire. It will be confirmed by reviewing their medical records.
Time Frame: 3 months
Population: Number of participants analyzed= 54 due to missing data. This question was displayed if answer to "Before this study, had you ever heard of PrEP?" was "Yes." Some participants obtained a PrEP prescription outside of the 3-month follow up timeframe (i.e., prior to their previous assessment), but did not fill their prescription at that time. These participants responded "No" to obtaining a PrEP prescription in the last 3-months, but "Yes" to filling their prescription in the last 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Number analyzed (Participants) | 26 | 28
Participants | 11 | 10
Statistical Analysis 1: Comparison: Patient Navigation (PN) vs Usual Care (UC); Test type: Superiority; p = .65, Regression, Logistic; Odds Ratio (OR) = 1.4

5. Primary Outcome: Percent of Participants That Initiated PrEP Use.
Description: Participants will be asked to self-report their PrEP initiation on a follow up questionnaire.
Time Frame: 3 months
Population: This question was displayed contingent on answering "Yes" to "Before this study, had you ever heard of PrEP?" Number of participants analyzed= 35. Some participants obtained and/or filled a PrEP prescription outside of the 3-month follow up timeframe (i.e., prior to their previous assessment), but did not initiate PrEP use at that time. These participants responded "No" to obtaining or filling a PrEP prescription in the last 3-months, but "Yes" to initiating PrEP in the last 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Number analyzed (Participants) | 18 | 17
Participants | 11 | 12
Statistical Analysis 1: Comparison: Patient Navigation (PN) vs Usual Care (UC); Test type: Superiority; p = .17, Regression, Logistic; Odds Ratio (OR) = .29

6. Primary Outcome: Percent of Participants That Adhered to PrEP Over the Past Seven Days for Participants That Initiated PrEP
Description: Participants will be asked to self-report their PrEP use over the past seven days on a follow up questionnaire.
Time Frame: 3 months
Population: This question was displayed if "Before this study, had you ever heard of PrEP?" was "Yes." Number of participants analyzed= 34. Some participants obtained and/or filled a PrEP prescription outside of the 3-month follow up timeframe (i.e., prior to their previous assessment), but did not initiate PrEP use at that time. These participants responded "No" to obtaining/filling a PrEP prescription in the last 3-months, but "Yes" to initiating PrEP in the last 3 months, and had adherence to report.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Number analyzed (Participants) | 18 | 16
Participants | 8 | 10
Statistical Analysis 1: Comparison: Patient Navigation (PN) vs Usual Care (UC); Test type: Superiority; p = .19, Regression, Logistic; Odds Ratio (OR) = .29

7. Primary Outcome: Percent of Participants That Attended PrEP Follow-up Appointment.
Description: Participants will be asked if they have attended a PrEP follow-up appointment on a follow up questionnaire. It will be confirmed by reviewing their medical records.
Time Frame: 3 months
Population: Data was not collected due to a coding error, thus the number of participants analyzed was zero.
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: March 12, 2020 through study completion, an average of 2 months
Description: A participant notified the study team that he was diagnosed with HIV and would like to discontinue participation in the study. The study team is uncertain of the exposure or diagnosis date. This information is Protected Health Information and the participant does not wish to continue participating, thus we will not have access to medical records for the exact date of the adverse event. All-cause mortality and other (not including serious) adverse events were not monitored/assessed.
Arm/Group | Patient Navigation (PN) | Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/29
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Navigation (PN) (N=28) | Usual Care (UC) (N=29)
Serious Adverse Event (Immune system disorders) | 0 (0) | 1 (1) — One participant in the usual care arm was diagnosed with HIV and chose to withdraw from study. The study team was notified on March 12, 2020 but the date of exposure and diagnosis is unknown, as that is protected health information.

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, all participant interactions were required to be virtual. The team was not able to obtain signed releases of information from PN-assigned participants during their final follow up assessment. Thus, it was not feasible to obtain supplementary medical records about PrEP cascade-related health information, as planned. Also, the team was not able to provide electronic MEMS cap devices to PrEP-prescribed participants to track adherence, as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT04048382/Prot_SAP_000.pdf